CLINICAL TRIAL: NCT06502132
Title: Comparison of the Effects of Therapeutic Touch and Patient Education on Postponed
Brief Title: Comparison of the Effects of Therapeutic Touch and Patient Education on Postponed Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Mehmet Gunay Uyar, Lecturer, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AtaturkU-SBE-MGU-01
Record Dates: First submitted 2024-07-05; First posted 2024-07-16 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Surgery
Keywords: surgery; postponement; anxiety; pain
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Intervention Model Description: Three groups with two experimental groups and one control group, including patient education and therapeutic touch
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control Group (No Intervention): Control group patients will receive routine care and no other intervention will be made within the scope of the study.
- Patient Education Group (Active Comparator): The patient education group will be informed about the waiting process that occurs as a result of surgery postponement through an education booklet prepared by the researcher in line with the literature.
  Interventions: Other: Patient Education Group
- Therapeutic Touch Group (Active Comparator): During the waiting period, patients will receive therapeutic touch by a certified researcher.
  Interventions: Other: Therapeutic Touch Group

INTERVENTIONS:
Other: Patient Education Group — Patients whose surgery has been postponed will be educated by the researcher through a booklet regarding the waiting process. The education includes information such as anxiety management, pain management, and re-surgery planning. The booklet consists of 22 pages and a copy is given to each patient in this group. The education lasts between 15-20 minutes and the patients' questions are answered. It is applied in a single session.
  Arms: Patient Education Group
Other: Therapeutic Touch Group — Therapeutic touch application is applied as a single session and lasts approximately 20-25 minutes. The therapeutic touch that emerges from the artistic aspect of nursing is an energybased practice that does not involve physical contact. Therapeutic touch is a conscious and compassionate effort to direct the flow of one's universal life energy to healing by influencing this energy.
  Arms: Therapeutic Touch Group

SUMMARY:
The aim of this study is to examine the effect of therapeutic touch and patient education on anxiety, pain, satisfaction levels and physiological parameters of patients and to determine patient experiences. The study will be conducted as a mixed method study. In the study, the effects of therapeutic touch and patient education on anxiety, satisfaction, pain levels and physiological parameters will be compared and the results will be compared. At the same time, qualitative statements of patients will be analyzed in depth and quantitative data will be supported.

DETAILED DESCRIPTION:
The study will be conducted with a nested design mixed method in which qualitative and quantitative methods will be used together with two experimental groups (education and therapeutic touch) and one control group. For the quantitative part, patients who meet the inclusion criteria will be randomized into the experimental and control groups. For randomization, two main groups will be formed as "major" and "minor" according to the degree of operation. The names of these two main groups will be written on two fans. Then both "major" and "minor" groups will be divided into "therapeutic touch group", "patient education group" and "control group". This separation will be done by writing the names of the subgroups on small pieces of paper, and when there is a patient whose surgery is postponed, after determining which main group the patient belongs to according to the degree of operation, a paper will be randomly drawn from the fan by the researcher, and the patient will be admitted to that group according to the subgroup name written on the paper. Only one of the patients lying in the same room will be included in the study to avoid interference. In addition, data will be collected from the patients assigned to all three groups as a result of randomization by using the phenomenological approach method, one of the qualitative research designs, using the face-to-face interview technique. In addition, data will be collected from the patients assigned to all three groups as a result of randomization by using face-to-face interview technique with the phenomenological approach method, one of the qualitative research designs. It is planned to collect qualitative and quantitative data from the same sample. Before collecting the data, the patients will be informed about the study, their written consent will be obtained verbally and digitally with the informed consent form, and then the 21-question Descriptive Characteristics Form will be applied as a conversation with verbal communication method. This process will contribute to the development of communication. Afterwards, the "State-Trait Anxiety Scale" will be applied to the patients in all groups, and qualitative data will be collected from the patients by applying the "Semi-structured Interview Form Before Interventions" prepared by the researcher in addition to the therapeutic touch and patient information groups. Afterwards, the relevant interventions (therapeutic touch or patient education) will be applied to the experimental groups. After the interventions are applied, the patients will be given one hour to rest. Afterwards, the state part of the "State-Trait Anxiety Scale", the "Numerical Proportioning Scale", the "Physiological Parameters Assessment Form" and the "Patient Satisfaction Assessment Form According to Watson Improvement Processes" will be applied to all groups as a post-test. In addition to the experimental groups, the "Semi-structured Interview Form After Interventions" prepared by the researcher will be administered.

Hypotheses of the Research:

H1: Patient education has a positive effect on anxiety in surgical patients whose operations have been postponed.

H2: Patient education has a positive effect on patient satisfaction in surgical patients whose operations have been postponed.

H3: Patient education has a positive effect on pain in surgical patients whose operations have been postponed.

H4: Patient education has a positive effect on physiological parameters in surgical patients whose operations have been postponed.

H5: Therapeutic touch has a positive effect on anxiety in surgical patients whose operations have been postponed.

H6: Therapeutic touch has a positive effect on patient satisfaction in surgical patients whose operations have been postponed.

H7: Therapeutic touch has a positive effect on pain in surgical patients whose operations have been postponed.

H8: Therapeutic touch has a positive effect on physiological parameters in surgical patients whose operations have been postponed Mixed Methods Research Question: How do the findings obtained through quantitative methods regarding the postponement process in surgical patients whose operations have been postponed correspond to the individual interview data conducted to explore the patients' feelings, thoughts, and experiences regarding the postponement process?

Qualitative Research Method Questions:

1) What are the feelings and thoughts of surgical patients whose operations have been postponed regarding the postponement situation? 2) What are the experiences of surgical patients whose operations have been postponed regarding the waiting process? 3) What is the relationship between the postponement of the operation and the anxiety, pain and satisfaction levels of the patients in surgical patients whose operations have been postponed? 4) What are the feelings and thoughts of surgical patients whose operations have been postponed regarding the interventions applied during the waiting process? 5) What are the experiences of surgical patients whose operations have been postponed regarding the interventions applied during the waiting process? 6) What are the expectations of surgical patients whose operations have been postponed from physicians and nurses during the waiting process? The study was planned to be conducted with 78 patients as a result of the power analysis test.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years of age or olde
* To undergo surgery
* Postponement of the operation for 24 hours
* Being able to read, write and communicate in Turkish
* Not having any vision, hearing or speech problems
* Volunteering to participate in the study

Exclusion Criteria:

* Being under 18 years of age
* Complete cancellation of the operation
* Postponing the operation for more than 24 hours
* Having vision, hearing or speech problems that prevent communication

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2024-07-03 (Actual); Primary Completion 2024-08-05 (Actual); Study Completion 2024-12-27 (Actual)

PRIMARY OUTCOMES:
State-Trait Anxiety Inventory (STAI-TX) | pre-test: 10 min;post-test: 5 min
  The 4-point Likert-type scale consists of two sections, each with 20 questions. The total score that can be obtained from the scale varies between 20 and 80, with a low average score indicating low anxiety and a high average score indicating high anxiety. There are ten reverse items in the State Anxiety Scale (1st, 2nd, 5th, 8th, 20th, 22nd, 25th, 26th, 19th and 20th), and seven reverse items in the Trait Anxiety Scale (21st, 26th, 37th, 30th, 33rd, 36th and 39th). The total score is calculated by subtracting the total weighted score of the reverse items from the total weighted score obtained for the direct items.

SECONDARY OUTCOMES:
Numeric Rating Scale (NRS) | Pre-test: Administered when the patient is informed about the postponement of the surgery (5 seconds for the patient to answer). Post-test: administered again 1 hour after the pre-test is completed (patient responds in 5 seconds).
  This scale, which is used to determine the intensity of pain, requires the patient to describe their pain in numbers. The NRS is a one-dimensional scale consisting of a horizontal line with the words "0 = No pain" on one side and "10 = Unbearable pain" on the other side to measure the level of pain. The score marked by the patient on the scale indicates the level of pain. The higher the marked score, the more severe the pain level becomes. The NRS has been proven to be a valid and reliable measurement tool in determining the intensity of acute pain after surgery in adult and elderly patients and is widely used in clinical and research areas.
Patient Satisfaction Evaluation Form According to Watson Improvement Processes | 5 min
  The first five questions consist of seven-point Likert-type questions scored between 1 and 7. "1" is never, "7" is always, and the sixth question is answered with "Yes-No." The seventh question consists of an open-ended question that evaluates the "moments of care application" in the applied nursing care.

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University Health Sciences Institute, Erzurum, Yakutiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No